CLINICAL TRIAL: NCT02686814
Title: A Multi-center, Non-randomized Trial to Determine the Safety and Effectiveness of the 17mm MDT-2215 Aortic Valve Bioprosthesis in Patients With Aortic Valve Disease
Brief Title: PERIGON Japan Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Surgery (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT-2215
Record Dates: First submitted 2015-12-15; First posted 2016-02-22 (Estimated); Results first posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2023-10

CONDITIONS: Aortic Stenosis
Keywords: Valvular heart disease; Severe aortic stenosis; Aortic valve replacement
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MDT-2215 (Experimental): 17mm MDT-2215 aortic valve bioprosthesis
  Interventions: Device: 17mm MDT-2215 aortic valve bioprosthesis

INTERVENTIONS:
Device: 17mm MDT-2215 aortic valve bioprosthesis

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the 17mm MDT-2215 aortic valve bioprosthesis.

DETAILED DESCRIPTION:
This is a prospective, interventional, non-randomized, multi-center trial, with each site following a common protocol in Japan. A maximum of 20 subjects will be implanted at a maximum of 10 sites in Japan. The trial will include male and female patients of legal age to provide informed consent in Japan, requiring replacement for a diseased, damaged, or malfunctioning native or prosthetic aortic valve. Patients will be followed and assessed after implant for up to 5 years.

This clinical trial information was submitted voluntarily under the applicable law and therefore, certain submission deadlines may not apply. (that is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CRF 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act of 42 CRF 11.24 and 11.44.)

ELIGIBILITY:
Inclusion Criteria:

1. Patient has severe aortic stenosis or regurgitation, and there is clinical indication for replacement of their native or prosthetic aortic valve with a bioprosthesis, with or without concomitant procedures, which are limited to any of the following:

   * Left atrial appendage (LAA) ligation
   * Coronary artery bypass graft (CABG)
   * Patent foramen ovale (PFO) closure
   * Ascending aortic aneurysm or dissection repair not requiring circulatory arrest
   * Resection of a sub-aortic membrane not requiring myectomy
2. Patient is geographically stable and willing to return to the implanting site for all follow-up visits
3. Patient is of legal age to provide informed consent
4. Patient has been adequately informed of risks and requirements of the trial and is willing and able to provide informed consent for participation in the clinical trial
5. In the opinion of the investigator, pre-operative imaging indicates the patient may be suitable for a 17mm size valve

Exclusion Criteria:

1. Patient has a pre-existing prosthetic valve or annuloplasty device in another position or requires replacement or repair of the mitral, pulmonary or tricuspid valve
2. Patient has had previous implant and then explant of the MDT-2215 aortic valve bioprosthesis
3. Patient presents with active endocarditis, active myocarditis or other systemic infection
4. Patient has an anatomical abnormality which would increase surgical risk of morbidity or mortality, including:

   * Ascending aortic aneurysm or dissection repair requiring circulatory arrest
   * Acute type A aortic dissection
   * Ventricular aneurysm
   * Porcelain aorta
   * Hostile mediastinum
   * Hypertrophic obstructive cardiomyopathy (HOCM)
   * Documented pulmonary hypertension (systolic >60mmHg)
5. Patient has a non-cardiac major or progressive disease, with a life expectancy of less than 2 years. These conditions include, but are not limited to:

   * Child-Pugh Class C liver disease
   * Terminal cancer
   * End-stage lung disease
6. Patient has renal failure, defined as dialysis therapy or glomerular filtration rate (GFR)<30 mL/min/1.73 m2
7. Patient has hyperparathyroidism
8. Patient is participating in another investigational device or drug trial or observational competitive study
9. Patient is pregnant, lactating or planning to become pregnant
10. Patient has a documented history of substance (drug or alcohol) abuse
11. Patient has greater than mild mitral valve regurgitation or greater than mild tricuspid valve regurgitation as assessed by echocardiography
12. Patient has systolic ejection fraction (EF)<20% as assessed by echocardiography
13. Patient has grade IV diastolic dysfunction
14. Patient has documented bleeding diatheses
15. Patient has had an acute preoperative neurological deficit or myocardial infarction and has not returned to baseline or stabilized ≥30 days prior to enrollment
16. Patient requires emergency surgery
17. Patient is in NYHA Class I
18. Operative Exclusion Criteria:

    * 1.) Prior to attempted implant of MDT-2215 valve, it is identified the patient requires a concomitant procedure not allow per the enrollment exclusion criteria
    * 2.) Patient anatomy is not suitable for implant of a size 17mm MDT-2215 aortic valve bioprosthesis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2022-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yutaka Okita, MD, Principal Investigator — Kobe University Hospital, Japan
Locations (10):
- Japan (10):
  - Chiba-Nishi General Hospital, Chiba
  - Kobe University Hospital, Hyogo Prefecture
  - Hyogo Prefectural Harima-Himeji General Medical Center, Hyogo Prefecture
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto
  - Kurashiki Central Hospital, Okayama
  - National Cerebral and Cardiovascular Center, Osaka
  - Saitama Medical Center, Jichi Medical University, Saitama
  - Saitama Medical University International Medical Center, Saitama
  - Tokushima Red Cross Hospital, Tokushima
  - Sakakibara Heart Institute, Tokyo

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MDT-2215
Started | 25
Completed | 6
Not Completed | 19
Not completed — Physician Decision | 14
Not completed — Withdrawal by Subject | 4
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Data from 11 participants implanted with MDT-2215 17mm valve from 25 enrolled participants
Arm/Group | MDT-2215
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.7 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline characteristics were summarized only on those implanted.
  Participants
    Hispanic or Latino | 0
    Not Hispanic or Latino | 11
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline characteristics were summarized only on those implanted.
  Participants
    American Indian or Alaska Native | 0
    Asian | 11
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 0
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Japan | 11
New York Heart Association (NYHA) Classification [Count of Participants; unit: Participants] — Cardiac Disease with Functional Classes I - No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation or shortness of breath.
  II - Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, shortness of breath or chest pain.
  III - Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, shortness of breath or chest pain.
  IV - Symptoms of heart failure at rest. Any physical activity causes further discomfort. Population: Baseline characteristics were summarized only on those implanted.
  Participants
    Class I | 0
    Class II | 11
    Class III | 0
    Class IV | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Changes in NYHA Classification From Baseline to 1 Year Post-procedure
Description: Change in New York Heart Association (NYHA) functional classification from baseline to 1 year post-procedure will be evaluated.
  Measure Description: Cardiac Disease with Functional Classes (lower value is more desirable than higher value) I - No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation or shortness of breath.
  II - Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, shortness of breath or chest pain.
  III - Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, shortness of breath or chest pain.
  IV - Symptoms of heart failure at rest. Any physical activity causes further discomfort.
Time Frame: This outcome will be identified from measurement at baseline and 1 year.
Measure: Count of Participants; unit: Participants
Arm/Group | MDT-2215
Number analyzed (Participants) | 11
Participants
  Improved 1 Class | 10
  No Change | 1

2. Primary Outcome: Effective Orifice Area Index at Baseline and 1 Year Post-procedure
Description: Effective Orifice Area Index (EOAI) at 1 year post-procedure will be evaluated. Effective Orifice Area Index (EOAI) in cm^2/m^2 EOAI = EOA/BSA Where: EOA is the effective orifice area in cm^2, and BSA is the body surface area in m^2
Time Frame: This outcome will be measured at 1 year.
Measure: Mean (Standard Deviation); unit: cm^2/m^2
Arm/Group | MDT-2215
Number analyzed (Participants) | 11
cm^2/m^2
  Baseline | 0.44 (0.14)
  1 Year | 0.82 (0.17)

3. Primary Outcome: Number of Participants With Composite New York Heart Association (NYHA) Classification and Effective Orifice EOAI Endpoint Improvement From Baseline to 1 Year
Description: Composite number of participants with NYHA change from baseline to 1 year post-procedure of 1 or greater and effective number of participants with effective EOAI 0.6cm^2/m^2 or greater at 1 year post implant will be evaluated. The objective is met if at least 60% of the subjects achieve the specified improvement in NYHA and EOAI.
  See Objective 1 for NYHA definition See Objective 2 for EOAI definition
Time Frame: This outcome will be identified from measurement at baseline and 1 year.
Measure: Count of Participants; unit: Participants
Arm/Group | MDT-2215
Number analyzed (Participants) | 11
Participants | 9

4. Secondary Outcome: Assessment of NYHA Functional Classification for Participants From Baseline up to 5 Years
Description: NYHA functional classification evaluation at baseline, discharge up to 30 days, 3-6 months, 1 year and annually thereafter up to 5 years.
  Measure Description: Cardiac Disease with Functional Classes I - No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation or shortness of breath.
  II - Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, shortness of breath or chest pain.
  III - Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, shortness of breath or chest pain.
  IV - Symptoms of heart failure at rest. Any physical activity causes further discomfort.
Time Frame: This outcome will be evaluated at baseline, discharge up to 30 days, 3-6 months, 1 year and annually thereafter up to 5 years.
Population: Subjects excited prior to visit. Year 2: 1 subject (death) Year 4: 1 subject (withdraw/other) Year 5: 3 subjects (withdraw/other)
Measure: Count of Participants; unit: Participants
Arm/Group | MDT-2215
Number analyzed (Participants) | 11
Participants
  Baseline: NYHA Classification I | 0
  Baseline: NYHA Classification II | 11
  Baseline: NYHA Classification III | 0
  Baseline: NYHA Classification IV | 0
  Baseline: NYHA Classification V | 0
  Baseline: Not done | 0
  Discharge up to 30 days: NYHA Classification I | 11
  Discharge up to 30 days: NYHA Classification II | 0
  Discharge up to 30 days: NYHA Classification III | 0
  Discharge up to 30 days: NYHA Classification IV | 0
  Discharge up to 30 days: NYHA Classification V | 0
  Discharge up to 30 days: Not done | 0
  3-6 Months: NYHA Classification I | 10
  3-6 Months: NYHA Classification II | 1
  3-6 Months: NYHA Classification III | 0
  3-6 Months: NYHA Classification IV | 0
  3-6 Months: NYHA Classification V | 0
  3-6 Months: Not done | 0
  1 Year: NYHA Classification I | 10
  1 Year: NYHA Classification II | 1
  1 Year: NYHA Classification III | 0
  1 Year: NYHA Classification IV | 0
  1 Year: NYHA Classification V | 0
  1 Year: Not done | 0
  2 Year: number analyzed (Participants) | 10
  2 Year: NYHA Classification I | 7
  2 Year: NYHA Classification II | 3
  2 Year: NYHA Classification III | 0
  2 Year: NYHA Classification IV | 0
  2 Year: NYHA Classification V | 0
  2 Year: Not done | 0
  3 Year: number analyzed (Participants) | 10
  3 Year: NYHA Classification I | 8
  3 Year: NYHA Classification II | 2
  3 Year: NYHA Classification III | 0
  3 Year: NYHA Classification IV | 0
  3 Year: NYHA Classification V | 0
  3 Year: Not done | 0
  4 Year: number analyzed (Participants) | 9
  4 Year: NYHA Classification I | 6
  4 Year: NYHA Classification II | 2
  4 Year: NYHA Classification III | 0
  4 Year: NYHA Classification IV | 0
  4 Year: NYHA Classification V | 0
  4 Year: Not done | 1
  5 Year: number analyzed (Participants) | 6
  5 Year: NYHA Classification I | 6
  5 Year: NYHA Classification II | 0
  5 Year: NYHA Classification III | 0
  5 Year: NYHA Classification IV | 0
  5 Year: NYHA Classification V | 0
  5 Year: Not done | 0

5. Secondary Outcome: Mean Effective Orifice Area Index (cm^2/m^2) From Baseline up to 5 Years
Description: Effective orifice area index at baseline, discharge up to 30 days, 3-6 months, 1 year and annually thereafter through 5 years as measured by effective orifice area (cm^2) per unit body surface area (m^2). The achievement criterion for the effective orifice area index (EOAI) is defined to be ≥0.6 cm^2/m^2.
  Effective Orifice Area Index (EOAI) in cm^2/m^2 EOAI = EOA/BSA Where: EOA is the effective orifice area in cm^2, and BSA is the body surface area in m^2
Time Frame: as for outcome 4
Population: Subject data for this outcome measure is limited by the number of subjects remaining in study at each timepoint and limited to those with non-missing measurements.
Measure: Mean (Standard Deviation); unit: cm^2/m^2
Arm/Group | MDT-2215
Number analyzed (Participants) | 11
cm^2/m^2
  Baseline: number analyzed (Participants) | 10
  Baseline | 0.44 (0.14)
  Discharge up to 30 days: number analyzed (Participants) | 10
  Discharge up to 30 days | 0.82 (0.16)
  3-6 Month | 0.77 (0.18)
  1 Year | 0.82 (0.17)
  2 Year: number analyzed (Participants) | 9
  2 Year | 0.70 (0.16)
  3 Year: number analyzed (Participants) | 9
  3 Year | 0.78 (0.16)
  4 Year: number analyzed (Participants) | 7
  4 Year | 0.76 (0.13)
  5 Year: number analyzed (Participants) | 5
  5 Year | 0.66 (0.16)

6. Secondary Outcome: Effective Orifice Area (cm^2) From Baseline up to 5 Years
Description: This will be measured by transthoracic echocardiography technique and will be assessed by an independent core laboratory.
Time Frame: This outcome will be evaluated at discharge up to 30 days, 3-6 months, 1 year and annually thereafter up to 5 years.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | MDT-2215
Number analyzed (Participants) | 11
cm^2
  Baseline: number analyzed (Participants) | 10
  Baseline | 0.58 (0.19)
  Discharge up to 30 Days: number analyzed (Participants) | 10
  Discharge up to 30 Days | 1.08 (0.19)
  3-6 Month | 1.03 (0.29)
  1 Year | 1.10 (0.22)
  2 Year: number analyzed (Participants) | 9
  2 Year | 0.96 (0.21)
  3 Year: number analyzed (Participants) | 9
  3 Year | 1.05 (0.23)
  4 Year: number analyzed (Participants) | 7
  4 Year | 1.04 (0.19)
  5 Year: number analyzed (Participants) | 5
  5 Year | 0.90 (0.21)

7. Secondary Outcome: Peak Pressure Gradient (mmHg) From Discharge up to 5 Years
Description: as for outcome 6
Time Frame: This outcome will be evaluated at discharge up to 30 days, 3-6 months, 1 year and annually thereafter up to 5 years.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MDT-2215
Number analyzed (Participants) | 11
mmHg
  Basline | 85.3 (29.7)
  Discharge up to 30 Days | 33.5 (11.0)
  3-6 Month | 36.5 (9.6)
  1 Year | 34.7 (12.7)
  2 Year: number analyzed (Participants) | 10
  2 Year | 35.6 (11.4)
  3 Year: number analyzed (Participants) | 10
  3 Year | 32.5 (11.1)
  4 Year: number analyzed (Participants) | 8
  4 Year | 33.4 (12.2)
  5 Year: number analyzed (Participants) | 5
  5 Year | 41.8 (9.0)

8. Secondary Outcome: Mean Pressure Gradient (mmHg) From Discharge up to 5 Years
Description: as for outcome 6
Time Frame: This outcome will be evaluated at discharge up to 30 days, 3-6 months, 1 year and annually thereafter up to 5 years.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MDT-2215
Number analyzed (Participants) | 11
mmHg
  Baseline | 53.3 (17.7)
  Discharge up to 30 Days | 18.5 (5.2)
  3-6 Month | 20.6 (5.8)
  1 Year | 20.9 (8.2)
  2 Year: number analyzed (Participants) | 10
  2 Year | 20.3 (5.7)
  3 Year: number analyzed (Participants) | 10
  3 Year | 18.8 (6.4)
  4 Year: number analyzed (Participants) | 8
  4 Year | 18.5 (6.5)
  5 Year: number analyzed (Participants) | 5
  5 Year | 24.2 (5.1)

9. Secondary Outcome: Degree of Paravalvular Regurgitation From Discharge up to 5 Years
Description: as for outcome 6
Time Frame: This outcome will be evaluated at discharge up to 30 days, 3-6 months, 1 year and annually thereafter up to 5 years.
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | MDT-2215
Number analyzed (Participants) | 11
Participants
  Discharge up to 30 Days: None | 8
  Discharge up to 30 Days: Trace | 1
  Discharge up to 30 Days: Mild | 1
  Discharge up to 30 Days: Moderate | 1
  Discharge up to 30 Days: Severe | 0
  Discharge up to 30 Days: Not Acquired | 0
  Discharge up to 30 Days: Not Evaluable | 0
  3-6 Months: None | 9
  3-6 Months: Trace | 0
  3-6 Months: Mild | 1
  3-6 Months: Moderate | 1
  3-6 Months: Severe | 0
  3-6 Months: Not Acquired | 0
  3-6 Months: Not Evaluable | 0
  1 Year: None | 10
  1 Year: Trace | 0
  1 Year: Mild | 0
  1 Year: Moderate | 1
  1 Year: Severe | 0
  1 Year: Not Acquired | 0
  1 Year: Not Evaluable | 0
  2 Year: number analyzed (Participants) | 10
  2 Year: None | 9
  2 Year: Trace | 0
  2 Year: Mild | 0
  2 Year: Moderate | 1
  2 Year: Severe | 0
  2 Year: Not Acquired | 0
  2 Year: Not Evaluable | 0
  3 Year: number analyzed (Participants) | 10
  3 Year: None | 9
  3 Year: Trace | 0
  3 Year: Mild | 0
  3 Year: Moderate | 1
  3 Year: Severe | 0
  3 Year: Not Acquired | 0
  3 Year: Not Evaluable | 0
  4 Year: number analyzed (Participants) | 8
  4 Year: None | 6
  4 Year: Trace | 1
  4 Year: Mild | 0
  4 Year: Moderate | 0
  4 Year: Severe | 1
  4 Year: Not Acquired | 0
  4 Year: Not Evaluable | 0
  5 Year: number analyzed (Participants) | 5
  5 Year: None | 4
  5 Year: Trace | 0
  5 Year: Mild | 0
  5 Year: Moderate | 0
  5 Year: Severe | 0
  5 Year: Not Acquired | 0
  5 Year: Not Evaluable | 1

10. Secondary Outcome: Degree of Transvalvular Regurgitation From Discharge up to 5 Years
Description: as for outcome 6
Time Frame: This outcome will be evaluated at discharge up to 30 days, 3-6 months, 1 year and annually thereafter up to 5 years.
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | MDT-2215
Number analyzed (Participants) | 11
Participants
  Baseline: None | 1
  Baseline: Trace | 0
  Baseline: Mild | 8
  Baseline: Moderate | 1
  Baseline: Severe | 1
  Baseline: Not Acquired | 0
  Baseline: Not Evaluable | 0
  Discharge up to 30 Days: None | 10
  Discharge up to 30 Days: Trace | 1
  Discharge up to 30 Days: Mild | 0
  Discharge up to 30 Days: Moderate | 0
  Discharge up to 30 Days: Severe | 0
  Discharge up to 30 Days: Not Acquired | 0
  Discharge up to 30 Days: Not Evaluable | 0
  3-6 Months: None | 9
  3-6 Months: Trace | 2
  3-6 Months: Mild | 0
  3-6 Months: Moderate | 0
  3-6 Months: Severe | 0
  3-6 Months: Not Acquired | 0
  3-6 Months: Not Evaluable | 0
  1 Year: None | 9
  1 Year: Trace | 1
  1 Year: Mild | 0
  1 Year: Moderate | 0
  1 Year: Severe | 0
  1 Year: Not Acquired | 0
  1 Year: Not Evaluable | 1
  2 Year: number analyzed (Participants) | 10
  2 Year: None | 9
  2 Year: Trace | 0
  2 Year: Mild | 1
  2 Year: Moderate | 0
  2 Year: Severe | 0
  2 Year: Not Acquired | 0
  2 Year: Not Evaluable | 0
  3 Year: number analyzed (Participants) | 10
  3 Year: None | 10
  3 Year: Trace | 0
  3 Year: Mild | 0
  3 Year: Moderate | 0
  3 Year: Severe | 0
  3 Year: Not Acquired | 0
  3 Year: Not Evaluable | 0
  4 Year: number analyzed (Participants) | 8
  4 Year: None | 6
  4 Year: Trace | 2
  4 Year: Mild | 0
  4 Year: Moderate | 0
  4 Year: Severe | 0
  4 Year: Not Acquired | 0
  4 Year: Not Evaluable | 0
  5 Year: number analyzed (Participants) | 5
  5 Year: None | 3
  5 Year: Trace | 1
  5 Year: Mild | 0
  5 Year: Moderate | 0
  5 Year: Severe | 0
  5 Year: Not Acquired | 0
  5 Year: Not Evaluable | 1

11. Secondary Outcome: Degree of Total Valvular Regurgitation From Discharge up to 5 Years
Description: as for outcome 6
Time Frame: This outcome will be evaluated at discharge up to 30 days, 3-6 months, 1 year and annually thereafter up to 5 years.
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | MDT-2215
Number analyzed (Participants) | 11
Participants
  Baseline: None | 1
  Baseline: Trace | 0
  Baseline: Mild | 7
  Baseline: Moderate | 1
  Baseline: Severe | 2
  Baseline: Not Acquired | 0
  Baseline: Not Evaluable | 0
  Discharge up to 30 Days: None | 7
  Discharge up to 30 Days: Trace | 2
  Discharge up to 30 Days: Mild | 1
  Discharge up to 30 Days: Moderate | 1
  Discharge up to 30 Days: Severe | 0
  Discharge up to 30 Days: Not Acquired | 0
  Discharge up to 30 Days: Not Evaluable | 0
  3-6 Month: None | 7
  3-6 Month: Trace | 2
  3-6 Month: Mild | 1
  3-6 Month: Moderate | 1
  3-6 Month: Severe | 0
  3-6 Month: Not Acquired | 0
  3-6 Month: Not Evaluable | 0
  1 Year: None | 9
  1 Year: Trace | 1
  1 Year: Mild | 0
  1 Year: Moderate | 1
  1 Year: Severe | 0
  1 Year: Not Acquired | 0
  1 Year: Not Evaluable | 0
  2 Year: number analyzed (Participants) | 10
  2 Year: None | 9
  2 Year: Trace | 0
  2 Year: Mild | 0
  2 Year: Moderate | 1
  2 Year: Severe | 0
  2 Year: Not Acquired | 0
  2 Year: Not Evaluable | 0
  3 Year: number analyzed (Participants) | 10
  3 Year: None | 9
  3 Year: Trace | 0
  3 Year: Mild | 0
  3 Year: Moderate | 1
  3 Year: Severe | 0
  3 Year: Not Acquired | 0
  3 Year: Not Evaluable | 0
  4 Year: number analyzed (Participants) | 8
  4 Year: None | 5
  4 Year: Trace | 2
  4 Year: Mild | 0
  4 Year: Moderate | 0
  4 Year: Severe | 1
  4 Year: Not Acquired | 0
  4 Year: Not Evaluable | 0
  5 Year: number analyzed (Participants) | 5
  5 Year: None | 3
  5 Year: Trace | 1
  5 Year: Mild | 0
  5 Year: Moderate | 0
  5 Year: Severe | 0
  5 Year: Not Acquired | 0
  5 Year: Not Evaluable | 1

12. Secondary Outcome: Performance Index (L/Min) From Discharge up to 5 Years
Description: as for outcome 6
Time Frame: This outcome will be evaluated at discharge up to 30 days, 3-6 months, 1 year and annually thereafter up to 5 years.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | MDT-2215
Number analyzed (Participants) | 11
L/min
  Baseline: number analyzed (Participants) | 10
  Baseline | 0.3 (0.1)
  Discharge up to 30 Days: number analyzed (Participants) | 10
  Discharge up to 30 Days | 0.6 (0.1)
  3-6 Month | 0.5 (0.2)
  1 Year | 0.6 (0.1)
  2 Year: number analyzed (Participants) | 9
  2 Year | 0.5 (0.1)
  3 Year: number analyzed (Participants) | 9
  3 Year | 0.6 (0.1)
  4 Year: number analyzed (Participants) | 7
  4 Year | 0.6 (0.1)
  5 Year: number analyzed (Participants) | 5
  5 Year | 0.5 (0.1)

13. Secondary Outcome: Cardiac Output (L/Min) From Discharge up to 5 Years
Description: as for outcome 6
Time Frame: This outcome will be evaluated at discharge up to 30 days, 3-6 months, 1 year and annually thereafter up to 5 years.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | MDT-2215
Number analyzed (Participants) | 11
L/min
  Baseline: number analyzed (Participants) | 10
  Baseline | 4.0 (1.3)
  Discharge up to 30 Days: number analyzed (Participants) | 10
  Discharge up to 30 Days | 4.0 (0.8)
  3-6 Month | 3.9 (0.8)
  1 Year | 4.4 (0.9)
  2 Year: number analyzed (Participants) | 9
  2 Year | 3.7 (0.9)
  3 Year: number analyzed (Participants) | 9
  3 Year | 3.8 (0.6)
  4 Year: number analyzed (Participants) | 7
  4 Year | 3.6 (0.9)
  5 Year: number analyzed (Participants) | 5
  5 Year | 4.3 (0.9)

14. Secondary Outcome: Cardiac Index (L/Min/m^2) From Discharge up to 5 Years
Description: as for outcome 6
Time Frame: This outcome will be evaluated at discharge up to 30 days, 3-6 months, 1 year and annually thereafter up to 5 years.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | MDT-2215
Number analyzed (Participants) | 11
L/min/m^2
  Baseline: number analyzed (Participants) | 10
  Baseline | 3.0 (0.9)
  Discharge up to 30 Days: number analyzed (Participants) | 10
  Discharge up to 30 Days | 3.0 (0.6)
  3-6 Months | 3.0 (0.5)
  1 Year | 3.3 (0.6)
  2 Year: number analyzed (Participants) | 9
  2 Year | 2.6 (0.6)
  3 Year: number analyzed (Participants) | 9
  3 Year | 2.8 (0.4)
  4 Year: number analyzed (Participants) | 7
  4 Year | 2.6 (0.7)
  5 Year: number analyzed (Participants) | 5
  5 Year | 3.2 (0.7)

15. Secondary Outcome: Safety:Valve-related Adverse Events
Description: The early (<=30days post-procedure), late (>30days post-procedure) and 1-year participant counts of the following valve-related adverse events will be evaluated:
  * thromboembolism
  * thrombosis
  * hemorrhage
  * paravalvular leak
  * endocarditis
  * hemolysis
  * structural valve deterioration
  * non-structural dysfunction
  * reintervention
  * explant
  * death
Time Frame: This outcome will be evaluated at discharge up to 30 days, 3-6 months, 1 year and annually thereafter up to 5 years.
Measure: Count of Participants; unit: Participants
Arm/Group | MDT-2215
Number analyzed (Participants) | 11
Participants
  Valve-Related Adverse Events | 0
  Valve Reinterventions / Explants | 0
  Valve-Related Deaths | 0
  Structural Valve Deterioration | 0

16. Secondary Outcome: Quality of Life Assessment - Physical Component Summary (Physical Functioning, Role-physical, Bodily Pain, General Health, Vitality)
Description: SF-36 Questionnaire Physical Component Summary (physical functioning, role-physical, bodily pain, general health, vitality) at baseline, 3-6 months, 1 year and annually thereafter through 5 years, where a higher score indicates a higher physical quality of life.
  Physical Component Summary Scale Lowest possible score: -7.28 Highest possible score: 52.71
Time Frame: This outcome will be evaluated at baseline, 3-6 months, 1 year and annually thereafter up to 5 years.
Population: Subject data for this outcome measure is limited by the number of subjects remaining in study at each timepoint and limited to those with non-missing measurements. No SF-36 quality of life assessment was collected at 5 years.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MDT-2215
Number analyzed (Participants) | 11
score on a scale
  Baseline | 37.4 (17.3)
  3-6 Month | 35.5 (15.7)
  1 Year | 39.2 (17.3)
  2 Year: number analyzed (Participants) | 10
  2 Year | 39.5 (13.2)
  3 Year: number analyzed (Participants) | 10
  3 Year | 26.6 (17.0)
  4 Year: number analyzed (Participants) | 2
  4 Year | 36.1 (21.4)
Statistical Analysis 1: Comparison: MDT-2215; 3-6 Month compared to Baseline; Test type: Equivalence — Each of the scales, for each follow-up time compared to baseline, the null hypothesis that the median paired difference is zero will be tested against the two-sided alternative that the median is not zero. Wilcoxon signed-rank test will be used; p = 0.7646, Wilcoxon signed-rank test; Median Difference (Final Values) = -0.9
Statistical Analysis 2: Comparison: MDT-2215; 1 Year compared to Baseline; Test type: Equivalence — [test comment as in outcome 16, analysis 1]; p = 0.8984, Wilcoxon signed-rank test; Median Difference (Final Values) = 3.9
Statistical Analysis 3: Comparison: MDT-2215; 2 Year compared to Baseline; Test type: Equivalence — [test comment as in outcome 16, analysis 1]; p = 0.8457, Wilcoxon signed-rank test; Median Difference (Final Values) = -0.0
Statistical Analysis 4: Comparison: MDT-2215; 3 Year compared to Baseline; Test type: Equivalence — [test comment as in outcome 16, analysis 1]; p = 0.1309, Wilcoxon signed-rank test; Median Difference (Final Values) = -7.7
Statistical Analysis 5: Comparison: MDT-2215; 4 Year compared to Baseline; Test type: Equivalence — [test comment as in outcome 16, analysis 1]; p = 0.5000, Wilcoxon signed-rank test; Median Difference (Final Values) = -15.2

17. Secondary Outcome: Quality of Life Assessment - Mental Component Summary (Social Functioning, Role-emotional, Mental Health)
Description: SF-36 Questionnaire Mental Component Summary (social functioning, role-emotional, mental health) at baseline, 3-6 months, 1 year and annually thereafter through 5 years, where a higher score indicates a higher quality of mental life.
  Lowest possible score: 31.63 Highest possible score: 66.69
Time Frame: This outcome will be evaluated at baseline, 3-6 months, 1 year and annually thereafter up to 5 years.
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MDT-2215
Number analyzed (Participants) | 11
score on a scale
  Baseline | 52.0 (6.1)
  3-6 Month | 55.2 (10.0)
  1 Year | 57.3 (9.9)
  2 Year: number analyzed (Participants) | 10
  2 Year | 57.9 (6.1)
  3 Year: number analyzed (Participants) | 10
  3 Year | 53.0 (8.7)
  4 Year: number analyzed (Participants) | 2
  4 Year | 53.5 (2.1)
Statistical Analysis 1: Comparison: MDT-2215; 3-6 Month compared to Baseline; Test type: Equivalence — [test comment as in outcome 16, analysis 1]; p = 0.2783, Wilcoxon signed-rank test; Median Difference (Final Values) = 1.5
Statistical Analysis 2: Comparison: MDT-2215; 1 Year compared to Baseline; Test type: Equivalence — [test comment as in outcome 16, analysis 1]; p = 0.0674, Wilcoxon signed-rank test; Median Difference (Final Values) = 6.4
Statistical Analysis 3: Comparison: MDT-2215; 2 Year compared to Baseline; Test type: Equivalence — [test comment as in outcome 16, analysis 1]; p = 0.0371, Wilcoxon signed-rank test; Median Difference (Final Values) = 6.4
Statistical Analysis 4: Comparison: MDT-2215; 3 Year compared to Baseline; Test type: Equivalence — [test comment as in outcome 16, analysis 1]; p = 0.6953, Wilcoxon signed-rank test; Median Difference (Final Values) = 0.8
Statistical Analysis 5: Comparison: MDT-2215; 4 Year compared to Baseline; Test type: Equivalence — [test comment as in outcome 16, analysis 1]; p > 0.9999, Wilcoxon signed-rank test; Median Difference (Final Values) = 1.0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline through study exit, up to 5 years.
Arm/Group | MDT-2215
All-Cause Mortality (participants affected / at risk) | 1/11
Serious Adverse Events (participants affected / at risk) | 2/11
Other Adverse Events (participants affected / at risk) | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MDT-2215 (N=11)
Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax and Pleural Effusions Nec (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MDT-2215 (N=11)
Anemias (Blood and lymphatic system disorders) | 1 (1) — Procedure-Related
Thrombocytopenias (Blood and lymphatic system disorders) | 1 (1) — Procedure-Related
Supraventricular Arrhythmias (Cardiac disorders) | 3 (3) — Procedure-Related
Ventricular Arrhythmias and Cardiac Arrest (Cardiac disorders) | 1 (1) — Procedure-Related
Coagulation and Bleeding Analyses (Investigations) | 1 (1) — Procedure-Related
Digestive Enzymes (Investigations) | 1 (1) — Procedure-Related
Hepatobiliary Function Diagnostic Procedures (Investigations) | 1 (1) — Procedure-Related
Protein Metabolism Disorders (Metabolism and nutrition disorders) | 1 (1) — Procedure-Related
Disturbances in Initiating and Maintaining Sleep (Psychiatric disorders) | 1 (1) — Procedure-Related
Conditions Associated with Abnormal Gas Exchange (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Procedure-Related
Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Procedure-Related
Pneumothorax and Pleural Effusions (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Procedure-Related
Vascular Hypertensive Disorders (Vascular disorders) | 1 (1) — Procedure-Related
Upper Respiratory Tract Infections (Infections and infestations) | 1 (1) — Procedure-Related
Supraventricular Arrhythmias (Cardiac disorders) | 1 (1) — Device - Related

LIMITATIONS AND CAVEATS:
Every effort was undertaken to minimize missing data. Unless otherwise specified in each objective, no statistical techniques were used to impute missing data for continuous or categorical outcomes. If a subject's data were missing for any reason, that subject was not included in that portion of the analysis. The number of subjects included in each analysis was reported so that the reader can assess the potential impact of missing data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-11-21): https://cdn.clinicaltrials.gov/large-docs/14/NCT02686814/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-29): https://cdn.clinicaltrials.gov/large-docs/14/NCT02686814/SAP_001.pdf